CLINICAL TRIAL: NCT05791383
Title: Managing Inpatient Neuropsychiatric Conditions Using Wearable Auricular Vagus Stimulation: The iWAVE Pilot Trial
Brief Title: taVNS on the Inpatient Psychiatric Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Xiaolong Peng, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 00120876
Record Dates: First submitted 2023-01-04; First posted 2023-03-30 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- transcutaneous auricular neurostimulation (low dose) (Experimental): All taVNS procedures will be conducted using the Spark Biomedical device. Electrodes will be placed on the left auricle and we will use stimulation parameters similar to ongoing taVNS work (25Hz, 500us pulse width) and a duty cycle of 1 minute on, 30 s off, repeated for 30 minutes. The low dose taVNS group will receive up to 3 treatments per day over the course of 3 days (for a total of up to 9 treatments).
  Interventions: Device: transcutaneous auricular neurostimulation
- transcutaneous auricular neurostimulation (high dose) (Experimental): All taVNS procedures will be conducted using the Spark Biomedical device. Electrodes will be placed on the left auricle and we will use stimulation parameters similar to ongoing taVNS work (25Hz, 500us pulse width) and a duty cycle of 1 minute on, 30 s off, repeated for 30 minutes. The high dose taVNS group will receive up to 9 treatments in a single day.
  Interventions: Device: transcutaneous auricular neurostimulation

INTERVENTIONS:
Device: transcutaneous auricular neurostimulation — All transcutaneous auricular neurostimulation procedures will be conducted using the Spark Biomedical device. We will use stimulation parameters similar to ongoing taVNS work (25Hz, 500us pulse width) and a duty cycle of 1 minute on, 30 s off, repeated for 30 minutes. taVNS sessions are considered complete after 30minutes. Subsequent taVNS sessions may be repeated no less than 30minutes after prior session completion. All subjects will begin with taVNS administered to the left auricle, however, if they begin to experience any irritation or discomfort of the left ear, study team staff will offer subjects the option to stop stimulation or switch stimulation to the right auricle.

SUMMARY:
This is a research study to find out if mental health symptoms in patients admitted to the Institute of Psychiatry are affected by a form of ear stimulation called transcutaneous auricular vagus nerve stimulation, or taVNS. Participants will receive ear stimulation during their inpatient treatment at the Institute of Psychiatry. Participants will be randomly assigned to either receive ear stimulation for 1 day (up to 9 treatments over the course of a single day) or 3 days (up to 3 treatments per day), and will have a 50:50 chance of being in either group (like the flip of a coin). Each treatment will last up to 30 minutes and there will be a break of at least 30 minutes in between treatments. The study team will ask participants to complete a group of questionnaires at the beginning and end of the study. In addition, there are several questionnaires that will be completed daily while participants are receiving ear stimulation. Participants in the 1 day stimulation group will also receive 2 days of follow up questionnaires after the initial day of stimulation. The questionnaires will ask questions about mental health symptoms that subjects may or may not be experiencing, including questions about mood, anxiety, and sleep. The ear stimulation treatments will not interfere with the care subjects are receiving from the medical team. In order to qualify for this study, participants must be actively receiving inpatient care at the MUSC Institute of Psychiatry.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 and up
* English speaking
* Admitted to 3 North's inpatient unit in MUSC's Institute of Psychiatry (IOP)
* Have the capacity and ability to provide one's own consent and sign the informed consent document
* Primary depression diagnosis

Exclusion Criteria:

* Facial or ear pain or recent ear trauma.
* Metal implant devices in the head, heart or neck.
* History of brain surgery.
* History of myocardial infarction or arrhythmia, bradycardia.
* Acute exacerbation of a chronic respiratory disorder or acute COVID-related symptoms.
* Active GI symptoms with a history of diabetes mellitus or history of gastroparesis secondary to diabetes mellitus.
* Personal or family history of seizure or epilepsy or personal use of medications that substantially reduce seizure threshold (e.g., olanzapine, chlorpromazine, lithium).
* Personal history of head injury, concussion, or self-report of moderate to severe traumatic brain injury.
* Individuals suffering from frequent/severe headaches.
* Individuals with a reported history of psychosis or mania, or individuals who are actively manic or psychotic.
* Individuals who are catatonic or otherwise unable to participate in the informed consent process.
* Moderate to severe alcohol or substance use disorder.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-03-24 (Actual); Study Completion 2024-03-24 (Actual)

PRIMARY OUTCOMES:
Side Effect and Adverse Event Report | 4 days
  Subjects will be monitored for adverse effects while receiving treatments.

SECONDARY OUTCOMES:
General Anxiety Disorder-7 (GAD-7) Scale | 4 days
  Subjects will conduct pre- and post- anxiety assessments to understand if stimulation improves neuropsychiatric condition. Higher GAD-7 scores indicate higher anxiety symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina Institute of Psychiatry, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Austelle CW, Cox SS, Connolly DJ, Baker Vogel B, Peng X, Wills K, Sutton F, Tucker KB, Ashley E, Manett A, Cortese B, Short EB, Badran BW. Accelerated Transcutaneous Auricular Vagus Nerve Stimulation for Inpatient Depression and Anxiety: The iWAVE Open Label Pilot Trial. Neuromodulation. 2025 Jun;28(4):672-681. doi: 10.1016/j.neurom.2025.02.003. Epub 2025 Mar 19. PMID 40117415